CLINICAL TRIAL: NCT00190775
Title: A Randomized, Double-Blind Comparison of Placebo and Atomoxetine Hydrochloride Given Once a Day in Adults With Attention-Deficit/Hyperactivity Disorder: With a Secondary Examination of Impact of Treatment on Family Functioning
Brief Title: A Randomized, Double-Blind Comparison of Placebo and Atomoxetine Hydrochloride Given Once a Day in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9043; B4Z-US-LYCW (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2010-10-21 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2010-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Experimental): Atomoxetine 40 milligrams (mg) once daily (QD) for 3 days followed by 80 mg QD for 11 days OR 40 mg QD for 7 days followed by 80 mg QD for 7 days, then 60/80/100 mg as determined by the investigator up to 24 weeks, orally
  Interventions: Drug: Atomoxetine Hydrochloride
- Placebo (Placebo Comparator): Placebo is administered once daily (QD), orally for 24 weeks. At the end of 24 weeks, the placebo arm is titrated to atomoxetine 40 mg QD for 3 days followed by 80 mg QD for 11 days OR 40 mg QD for 7 days followed by 80 mg QD for 7 days, then 40-100 mg QD, orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride — Atomoxetine 40 mg QD for 3 days followed by 80 mg QD for 11 days OR 40 mg QD for 7 days followed by 80 mg QD for 7 days, then 60/80/100 mg as determined by the investigator up to 24 weeks, orally
  Other Names: LY139603; Strattera
  Arms: Atomoxetine
Drug: Placebo — Placebo is administered QD, orally for 24 weeks. At the end of 24 weeks, the placebo arm is titrated to atomoxetine 40 mg QD for 3 days followed by 80 mg QD for 11 days OR 40 mg QD for 7 days followed by 80 mg QD for 7 days, then 40-100 mg QD, orally.
  Arms: Placebo

SUMMARY:
This is a parallel design, double-blind, placebo-controlled, multi-center, 38-week treatment trial of atomoxetine in adults with attention deficit hyperactivity disorder (ADHD) who are currently living in a family situation with at least one child. The primary objective of the study is to demonstrate the efficacy of atomoxetine compared to placebo in the reduction of ADHD symptoms over 12 and 24 weeks of blinded treatment.

DETAILED DESCRIPTION:
The initial study was 34 weeks long; however, the protocol was amended to extend the open-label period of the study from 8 weeks to 12 weeks (38 weeks total).

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders Fourth Edition - Text Revision (DSM-IV-TR) criteria for Adult Attention-Deficit/Hyperactivity Disorder (ADHD) as assessed by the Conners' Adult ADHD Diagnostic Interview for DSM-IV (CAADID).
* Have a Clinical Global Impression for ADHD Severity Score (CGI-ADHD-S) of 4 or greater Visit 2 and 3.
* Adult Men and Women age 18 years or older at time informed consent is obtained.
* Must be in a reciprocal relationship with a person of the opposite sex living in same defined household (cohabitating) with their spouse/significant other for a period of at least 3 months. This spouse/significant other cannot change during the study.
* Must have one or more children 6-17 years of age living the home as the primary residence.

Exclusion Criteria:

* Anyone meeting Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria for any history of bipolar disorder or any history of a psychotic disorder.
* Anyone meeting diagnostic (DSM-IV) criteria for current major depression or current anxiety disorder.
* Taking psychotropic medications on a regular basis.
* Having any medical condition that would be exacerbated or not appropriate for inclusion in this trial.
* Previously taken an adequate trial of atomoxetine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2004-09; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (20):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irvine, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Libertyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bardstown, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester Hills, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troy, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Kisco, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Media, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Herndon, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleton, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Allis, Wisconsin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce, Puerto Rico

REFERENCES:
- [Result] Young JL, Sarkis E, Qiao M, Wietecha L. Once-daily treatment with atomoxetine in adults with attention-deficit/hyperactivity disorder: a 24-week, randomized, double-blind, placebo-controlled trial. Clin Neuropharmacol. 2011 Mar-Apr;34(2):51-60. doi: 10.1097/WNF.0b013e31820c00eb. PMID 21406998
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647

RESULTS

PARTICIPANT FLOW:
Groups:
- Atomoxetine: Atomoxetine 40 milligrams (mg) once daily (QD) for 3 days followed by 80 mg QD for 11 days OR 40 mg QD for 7 days followed by 80 mg QD for 7 days then 60/80/100 mg as determined by the investigator up to 24 weeks, orally
Period: Overall Study
Arm/Group | Atomoxetine | Placebo
Started | 268 | 234
Received Study Drug | 266 | 234
Completed | 119 | 134
Not Completed | 149 | 100
Not completed — Adverse Event | 57 | 22
Not completed — Satisfactory Response | 1 | 0
Not completed — Lack of Efficacy | 28 | 32
Not completed — Lost to Follow-up | 31 | 23
Not completed — Participant Moved | 0 | 1
Not completed — Withdrawal by Subject | 24 | 13
Not completed — Sponsor Decision | 1 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Noncompliance | 3 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Exclusion Criteria Met | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 268 | 234 | 502
Age Continuous [Mean (Standard Deviation); unit: Years] | 41.21 (6.89) | 41.39 (7.49) | 41.30 (7.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 132 | 263
  Male | 137 | 102 | 239
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic | 24 | 20 | 44
  Caucasian | 227 | 199 | 426
  African Descent | 11 | 6 | 17
  East/Southeast Asian | 0 | 2 | 2
  Western Asian | 1 | 0 | 1
  Other | 5 | 7 | 12
Region of Enrollment [Number; unit: Participants]
  United States | 255 | 224 | 479
  Puerto Rico | 13 | 10 | 23
Attention Deficit Hyperactivity Disorder (ADHD) Subtype [Number; unit: Participants]
  Combined | 179 | 166 | 345
  Inattentive | 89 | 67 | 156
  Hyperactive/Impulsive | 0 | 1 | 1
Previous Stimulant Exposure [Number; unit: Participants]
  Yes | 47 | 35 | 82
  No | 220 | 198 | 418
  Unknown or Not Reported | 1 | 1 | 2
Adult Attention Deficit Hyperactivity Disorder (ADHD) Investigator Symptom Rating Scale (AISRS) [Mean (Standard Deviation); unit: Units on a scale] — 18-item scale that captures the 18-item Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) symptoms of ADHD. 9 inattentive items alternate with 9 hyperactive/impulsive items. Each item is scored 0 (none), 1 (mild), 2 (moderate), or 3 (severe). The total score range is 0-54 (0-27 for each subscale). Higher scores indicate more impaired participants. The scale was administered by a physician or PhD at the investigative site.
  Units on a scale
    AISRS Total Score | 36.07 (7.64) | 36.59 (8.34) | 36.31 (7.97)
    AISRS Inattention Score | 20.91 (3.83) | 20.62 (4.02) | 20.77 (3.92)
    AISRS Hyperactivity Score | 15.16 (5.75) | 15.97 (5.94) | 15.54 (5.85)
Alabama Parenting Questionnaire (APQ) [Mean (Standard Deviation); unit: Units on a scale] — 42-item scale, 3 subscales (z-scores [-2 to 2]): Dysfunctional/Negative/Positive Parenting. Each construct rated 1=never/5=always (# items): involvement (10), supervision (10), positive parenting (6), inconsistent discipline (6), other discipline (7), harsh discipline (3). Higher scores indicate impairment: dysfunctional/negative parenting composite; supervision, inconsistent discipline, harsh punishment, other discipline. Lower scores indicate impairment: positive parenting composite; positive parenting, involvement. Completed by participants with a child 6-12 or 13-17 years living at home.
  Units on a scale
    Child Involvement Mother | 35.30 (6.02) | 36.09 (5.90) | 35.67 (5.97)
    Child Involvement Father | 31.50 (6.85) | 32.35 (6.86) | 31.90 (6.86)
    Child Positive Parenting | 23.85 (4.04) | 23.40 (4.02) | 23.64 (4.03)
    Child Poor Monitoring/Supervision | 16.93 (4.92) | 17.27 (5.34) | 17.09 (5.12)
    Child Inconsistent Discipline | 12.66 (3.44) | 13.01 (3.57) | 12.83 (3.50)
    Child Corporal Punishment | 4.86 (2.08) | 4.99 (2.37) | 4.92 (2.22)
    Child Other Discipline Practice | 17.62 (3.52) | 18.18 (3.88) | 17.88 (3.70)
    Parent Involvement | 37.71 (5.11) | 37.61 (5.62) | 37.67 (5.34)
    Parent Positive Parenting | 24.53 (3.26) | 24.06 (3.58) | 24.31 (3.42)
    Parent Poor Monitoring Supervision | 16.64 (4.91) | 16.50 (4.78) | 16.58 (4.85)
    Parent Inconsistent Discipline | 15.37 (3.44) | 15.48 (3.42) | 15.42 (3.42)
    Parent Corporal Punishment | 4.73 (1.60) | 4.75 (1.76) | 4.74 (1.67)
    Parent Other Discipline Practice | 19.53 (3.08) | 19.64 (2.96) | 19.58 (3.02)
    Parent Dysfunctional Parenting Composite | 0.12 (0.98) | 0.17 (1.01) | 0.14 (0.99)
    Parent Negative Parenting | 0.21 (1.05) | 0.21 (0.99) | 0.21 (1.02)
    Parent Positive Parenting | -0.00 (0.95) | -0.07 (1.05) | -0.04 (1.00)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms/square meters] — Body mass index (BMI) is an estimate of body fat based on body weight divided by height squared.
  Kilograms/square meters | 30.15 (6.58) | 29.31 (6.51) | 29.76 (6.56)
Child Disruptive Behavior Rating Scale (CDBRS) Parent Form [Mean (Standard Deviation); unit: Units on a scale] — Child Disruptive Behavior Rating Scale (CDBRS) contains the symptoms of ADHD (9 items for Inattention/9 items for Hyperactive-Impulsive). Total maximum severity score is 54 (0-27 for each subscore). Higher scores indicate greater impairment. Participants with a child aged 6-12 or 13-17 years old living in the home completed the scale.
  Units on a scale
    Total Score | 24.56 (13.30) | 24.35 (13.01) | 24.46 (13.16)
    Inattention Symptom ADHD Score | 13.39 (7.30) | 13.35 (6.86) | 13.37 (7.09)
    Hyperactive-Impulsive Symptom ADHD Score | 11.17 (6.98) | 11.00 (6.95) | 11.09 (6.96)
Clinical Global Improvement Attention Deficit Hyperactivity Disorder Severity (CGI-ADHD-S) [Mean (Standard Deviation); unit: Units on a scale] — The CGI-ADHD-S is a single-item rating of the clinician's assessment of the severity of ADHD symptoms in relation to the clinician's total experience with ADHD subjects. Severity is rated on a 7-point scale (1=normal, not at all ill; 7=among the most extremely ill subjects). The scale was administered by a physician or PhD at the investigative site.
  Units on a scale | 4.56 (0.62) | 4.58 (0.60) | 4.57 (0.61)
Conners' Adult ADHD Rating Scale Screening Version (CAARS-Inv:SV) [Mean (Standard Deviation); unit: Units on a scale] — 30-item scale containing 3 subscales: inattention (9 items), hyperactivity/ impulsivity (9 items), and ADHD Index (12 items). Each item is scored 0-3 (0=not at all/never; 1=just a little/once in a while; 2=pretty much/often; 3=very much/very frequently). Total ADHD symptoms score=sum of the inattention and hyperactivity/impulsivity subscales. Total Scores range from 0-54 (range of 0-27 for the inattention and hyperactivity subscales; 0-36 for the ADHD Index) with higher scores indicating more impaired participants. The scale was administered by a physician/PhD at the investigative site.
  Units on a scale
    Total ADHD Symptoms Score | 34.64 (8.39) | 35.50 (8.53) | 35.04 (8.46)
    Inattention Subscale | 19.97 (4.45) | 19.90 (4.33) | 19.94 (4.39)
    Hyper/Impulsive Subscale | 14.67 (5.89) | 15.60 (5.80) | 15.11 (5.86)
    Index Subscale | 21.60 (5.37) | 21.49 (5.74) | 21.55 (5.54)
Dyadic Adjustment Scale (DAS) - Participant (Self) [Mean (Standard Deviation); unit: T-scores of units on a scale] — 32-item self-report scale to assess quality of the relationship perceived by participants. Response anchors vary and include a 5-, 6- or 7-point Likert scale (always agree/disagree; all the time/never); and 2 yes/no items. Assesses 4 relationship aspects (# items): dyadic satisfaction (10), cohesion (5), and consensus (13), affectional expression (4). Raw score total=0-151 and is converted to a t-score (0-100; mean=50, standard deviation (SD)=10). T-scores of 45-55 indicate a typical score (no concern). Scores <30 indicate significant impairment. Lower scores indicate poorer dyadic adjustment.
  T-scores of units on a scale
    Total Dyadic Adjustment | 43.06 (11.90) | 42.37 (11.11) | 42.74 (11.53)
    Affectional Expression | 43.70 (12.52) | 44.85 (11.68) | 44.24 (12.14)
    Dyadic Cohesion | 52.51 (10.63) | 51.58 (10.02) | 52.08 (10.35)
    Dyadic Consensus | 44.99 (9.22) | 44.26 (8.69) | 44.65 (8.98)
    Dyadic Satisfaction | 42.98 (10.82) | 42.49 (10.24) | 42.75 (10.55)
Dyadic Adjustment Scale (DAS) - Spouse/Significant Other [Mean (Standard Deviation); unit: T-scores of units on a scale] — 32-item self-report scale to assess quality of the relationship perceived by the spouse/significant other. Response anchors vary and include a 5-, 6- or 7-point Likert scale (always agree/disagree; all the time/never); and 2 yes/no items. Assesses 4 relationship aspects (# items): dyadic satisfaction (10), cohesion (5), and consensus (13), and affectional expression (4). Raw score total=0-151 and is converted to a t-score (0-100; mean=50, SD=10). T-scores of 45-55 indicate a typical score (no concern). Scores <30 indicate significant impairment. Lower scores indicate poorer dyadic adjustment.
  T-scores of units on a scale
    Total Dyadic Adjustment | 41.93 (11.44) | 41.75 (11.29) | 41.85 (11.36)
    Affectational Expression | 43.18 (11.97) | 43.66 (12.28) | 43.41 (12.10)
    Dyadic Cohesion | 51.35 (11.09) | 51.70 (10.30) | 51.51 (10.72)
    Dyadic Consensus | 40.82 (10.18) | 40.44 (10.02) | 40.64 (10.10)
    Dyadic Satisfaction | 42.25 (10.75) | 41.84 (10.53) | 42.06 (10.64)
Family Assessment Measure III (FAM) Dyadic Relationship Scale (DRS) - Participant (Self) [Mean (Standard Deviation); unit: T-scores of units on a scale] — FAM consists of 3 components: General Scale; Dyadic Relationships Scale (DRS), and Self-Rating Scale. Participants completed the DRS scale, a 42-item self-report scale providing quantitative indices of family strengths/weaknesses. Items are rated 0-3 (strongly agree, agree, disagree, strongly disagree). Raw scores=0-18 (each subscale) and are converted to a t-score (mean=50, standard deviation=10; scores range from 0-100). T-scores should be between 40-60. T-scores >=60 indicate disturbance in family functioning.
  T-scores of units on a scale
    Task Accomplishment | 62.78 (5.56) | 62.38 (5.43) | 62.59 (5.50)
    Role Performance | 60.81 (5.03) | 61.13 (5.75) | 60.96 (5.37)
    Communication | 64.97 (6.49) | 64.24 (6.35) | 64.63 (6.43)
    Affective Expression | 61.48 (8.63) | 61.71 (9.47) | 61.59 (9.02)
    Involvement | 64.07 (7.92) | 64.59 (7.35) | 64.31 (7.66)
    Control | 62.70 (5.95) | 62.13 (6.07) | 62.43 (6.01)
    Values and Norms | 65.66 (6.70) | 64.90 (7.44) | 65.30 (7.06)
Family Assessment Measure III (FAM) Dyadic Relationship Scale (DRS) - Spouse/Significant Other [Mean (Standard Deviation); unit: T-scores of units on a scale] — FAM consists of 3 components: General Scale; Dyadic Relationships Scale (DRS), and Self-Rating Scale. The spouse/significant other completed the DRS scale, a 42-item self-report scale providing quantitative indices of family strengths/weaknesses. Items are rated 0-3 (strongly agree, agree, disagree, strongly disagree). Raw scores=0-18 (each subscale) and are converted to a t-score (mean=50, standard deviation (SD)=10; scores range from 0-100). T-scores should be between 40-60. T-scores >=60 indicate disturbance in family functioning.
  T-scores of units on a scale
    Task Accomplishment | 61.52 (5.97) | 60.90 (5.83) | 61.23 (5.91)
    Role Performance | 61.28 (5.67) | 60.59 (6.00) | 60.96 (5.83)
    Communication | 64.05 (6.37) | 63.47 (7.02) | 63.78 (6.68)
    Affective Expression | 61.97 (9.67) | 61.68 (9.07) | 61.84 (9.39)
    Involvement | 64.96 (8.95) | 64.52 (8.77) | 64.76 (8.86)
    Control | 61.98 (6.52) | 61.34 (6.25) | 61.68 (6.40)
    Values and Norms | 65.32 (7.11) | 65.52 (7.17) | 65.41 (7.13)
Height [Mean (Standard Deviation); unit: Centimeters] | 171.23 (10.37) | 170.01 (9.74) | 170.66 (10.09)
Montgomery-Asberg Depression Rating Scale Total Score (MADRS) [Mean (Standard Deviation); unit: Units on a scale] — The MADRS is an investigator administered rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
  Units on a scale | 8.13 (4.80) | 8.12 (5.01) | 8.13 (4.89)
Parent Stress Index (PSI) Total Stress and Life Stress [Mean (Standard Deviation); unit: Units on a scale] — The PSI 19-item Stress Life Events scale has yes/no responses and measures situational circumstances beyond control (death of family member, divorce, etc.) in the past 12 months. Maximum score (all answers=yes) is 79; a Life Stress raw score >=17 indicates high stress. Each question is weighted based upon the event. Total Score measures relative magnitude of stress in parent-child system. High scores (>=85th percentile) indicate higher stress. Total Stress >=258 is indicative of impairment. Participants with a child aged 6-12 or 13-17 years living at home completed the scale.
  Units on a scale
    Total Stress | 285.40 (53.45) | 277.11 (52.65) | 281.53 (53.18)
    Life Stress | 1.57 (3.56) | 1.76 (3.68) | 1.66 (3.62)
Parent Stress Index (PSI) Parent Domains [Mean (Standard Deviation); unit: Units on a scale] — 120-item scale includes 101 items rated on 5-point Likert scale (strongly agree/strongly disagree) or 4-5 point multiple choices. Adult Domain characteristics' subscales and score ranges include: Competence (13-65), Isolation (6-30), Attachment (7-35), Health (5-25), Role Restriction (7-35), Depression (9-45), Spouse (7-35). Total Score measures relative magnitude of stress in parent-child system. Parent Domain score >=148 (>=85th percentile) is indicative of impairment. Participants with a child aged 6-12 or 13-17 years living at home completed the scale.
  Units on a scale
    Parent Domain Total | 135.40 (25.22) | 130.22 (24.62) | 132.98 (25.05)
    Parent Domain Role Restriction | 18.93 (5.33) | 18.26 (4.99) | 18.62 (5.18)
    Parent Domain Depression | 22.79 (6.10) | 21.01 (5.68) | 21.96 (5.97)
    Parent Domain Spouse | 18.19 (5.03) | 18.14 (5.04) | 18.17 (5.03)
    Parent Domain Competence | 32.63 (6.69) | 31.78 (7.10) | 32.23 (6.89)
    Parent Domain Isolation | 15.49 (4.71) | 14.56 (4.61) | 15.06 (4.68)
    Parent Domain Attachment | 13.74 (4.21) | 12.95 (3.61) | 13.37 (3.96)
    Parent Domain Health | 13.72 (2.71) | 13.52 (2.62) | 13.63 (2.67)
Parent Stress Index (PSI) Child Domains [Mean (Standard Deviation); unit: Units on a scale] — 120-item scale includes 101 items rated on 5-point Likert scale (strongly agree/strongly disagree) or 4-5 point multiple choices. Child Domain characteristics' subscales and score ranges include: Distractibility/Hyperactivity (9-45), Adaptability (11-55), Reinforces Parent (6-30), Demandingness (9-45), Mood (5-25), Acceptability (7-35). Total Score measures relative magnitude of stress in parent-child system. A Child Domain score >=116 (>=85th percentile) is indicative of impairment. Participants with a child aged 6-12 or 13-17 years living at home completed the scale.
  Units on a scale
    Child Domain Total | 150.00 (34.46) | 146.88 (34.44) | 148.54 (34.45)
    Child Domain Distractibility/Hyperactivity | 27.49 (6.46) | 27.59 (6.48) | 27.54 (6.47)
    Child Domain Adaptability | 48.29 (11.56) | 47.59 (12.28) | 47.96 (11.89)
    Child Domain Reinforces Parent | 24.87 (7.13) | 23.75 (7.07) | 24.34 (7.12)
    Child Domain Demandingness | 20.99 (6.09) | 20.71 (6.48) | 20.85 (6.27)
    Child Domain Mood | 12.42 (3.89) | 12.06 (4.03) | 12.25 (3.96)
    Child Domain Acceptability | 15.94 (4.75) | 15.18 (4.67) | 15.59 (4.72)
Parenting Sense of Competence (PSOC) Scale [Mean (Standard Deviation); unit: Units on a scale] — 16-item scale to assess parenting self-esteem: the Satisfaction Subscale has 9 questions (2,3,4,5,8,9,12,14,16)=54; the Efficacy Subscale has 7 questions (1,6,7,10,11,13,15)=43. Each response on the satisfaction subscale is answered on a 6-point scale (strongly agree/strongly disagree). Higher scores indicate greater satisfaction and greater self-efficacy. Lower scores mean more impairment. Participants with a child aged 6-12 or 13-17 years living at home completed the scale.
  Units on a scale
    Total | 58.64 (9.83) | 60.80 (9.18) | 59.65 (9.58)
    Satisfaction Scale | 33.46 (6.58) | 34.94 (6.38) | 34.15 (6.52)
    Efficacy Scale | 25.18 (4.72) | 25.86 (4.31) | 25.50 (4.54)
State-Trait Anxiety Inventories (STAI) [Mean (Standard Deviation); unit: Units on a scale] — Self-report scale completed by the participant. Separate scales measure state (20 items) and trait (20 items) anxiety. The participant reports how they feel "right now at this moment" for state anxiety and how they "generally" feel for trait anxiety. The "state" items are scored as: 1 (not at all), 2 (somewhat true), 3 (moderately true), 4 (very true). The "trait" items are scored as: 1 (almost never), 2 (sometimes), 3 (often), 4 (almost always). Scores range from 4-80 for each scale. Higher scores indicate more impaired participants.
  Units on a scale
    State Anxiety Score | 40.13 (11.55) | 41.16 (11.18) | 40.61 (11.38)
    Trait Anxiety Score | 47.44 (10.68) | 46.05 (11.22) | 46.79 (10.94)
Weight [Mean (Standard Deviation); unit: Kilograms] | 88.22 (20.40) | 84.84 (19.72) | 86.65 (20.14)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24 Weeks in the Conners' Adult Attention Deficit Hyperactivity Disorder Rating Scale - Investigator Rated: Screening Version (CAARS-Inv:SV) Total ADHD Symptoms Score
Description: 30-item scale containing 3 subscales: inattention (9 items), hyperactivity/ impulsivity (9 items), and ADHD Index (12 items). Each item is scored 0-3 (0=not at all/never; 1=just a little/once in a while; 2=pretty much/often; 3=very much/very frequently). Total ADHD symptoms score=sum of the inattention and hyperactivity/impulsivity subscales. Total Scores range from 0-54 (range of 0-27 for the inattention and hyperactivity subscales; 0-36 for the ADHD Index) with higher scores indicating more impaired participants. The scale was administered by a physician/PhD at the investigative site.
Time Frame: Baseline, 24 weeks
Population: Participants with a baseline and at least one post-baseline CAARS Total ADHD Symptoms Score were included.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 125 | 136
Units on a scale | -16.43 (0.88) | -8.65 (0.85)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Approximately 500 participants were randomized to atomoxetine or placebo (1:1) which provided at least 90% power to detect a treatment difference of 3.64 points on the CAARS-Inv:SV Total ADHD Symptoms Score assuming a SD of 9.85 based on 2-sided significance level of 0.05 using a 2-sample t-test. Mean and SD assumptions were associated with effect size of 0.37 and 30% missing data rate. These assumptions applied to Weeks 12 and 24 treatment effects. Marginal power at Weeks 12 and 24 was 86%; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Model included visit, baseline, treatment, pooled investigator, child with ADHD, and treatment by visit; Mean Difference (Final Values) = -7.78, Standard Error of Mean 1.11 — Least Squares Mean Difference = Atomoxetine - Placebo

2. Secondary Outcome: Change From Baseline to 8 Weeks in the Family Assessment Measure Version III (FAM) Dyadic Relationship Scale (DRS) - Participant
Description: FAM consists of 3 components: General Scale; Dyadic Relationships Scale (DRS), and Self-Rating Scale. Participants completed the DRS scale, a 42-item self-report scale providing quantitative indices of family strengths/weaknesses. Items are rated 0-3 (strongly agree, agree, disagree, strongly disagree). Raw scores=0-18 (each subscale) and are converted to a t-score (mean=50, standard deviation (SD)=10; scores range from 0-100). T-scores should be between 40-60. T-scores >=60 indicate disturbance in family functioning.
Time Frame: Baseline, 8 weeks
Population: Intent-to-treat (ITT) population: participants were included in the ITT population if they had a baseline and at least one post-baseline efficacy measurement. Last observation carried forward (LOCF) was used.
Measure: Mean (Standard Deviation); unit: T-scores of units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
T-scores of units on a scale
  Task Accomplishment | -0.79 (6.66) | -0.41 (6.37)
  Role Performance | -0.25 (5.30) | -0.04 (6.18)
  Communication | -0.63 (7.50) | -0.29 (6.88)
  Affective Expression | 0.50 (7.75) | -0.33 (7.86)
  Involvement | -0.27 (7.79) | 0.17 (7.54)
  Control | -0.01 (6.64) | 0.33 (6.56)
  Values and Norms | 0.00 (6.97) | -0.27 (8.02)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.905, ANCOVA — P-Value for Task Accomplishment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.491, ANCOVA — P-Value for Role Performance; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.600, ANCOVA — P-Value for Communication; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.052, ANCOVA — P-Value for Affective Expression; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.514, ANCOVA — P-Value for Involvement; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.515, ANCOVA — P-Value for Control; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.315, ANCOVA — P-Value for Values and Norms; Model included treatment, pooled investigator, child with ADHD, and baseline

3. Secondary Outcome: Change From Baseline to 24 Weeks in the Family Assessment Measure Version III (FAM) Dyadic Relationship Scale (DRS) - Participant
Description: as for outcome 2
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-scores of units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
T-scores of units on a scale
  Task Accomplishment | -0.81 (6.45) | -0.90 (6.59)
  Role Performance | -0.33 (5.60) | 0.27 (6.65)
  Communication | -1.15 (7.49) | -0.58 (6.73)
  Affective Expression | 0.05 (8.31) | 0.25 (8.10)
  Involvement | -0.32 (7.68) | 0.56 (7.32)
  Control | -0.53 (6.89) | 0.41 (6.21)
  Values and Norms | -0.67 (7.15) | 0.31 (8.21)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.176, ANCOVA — P-Value for Task Accomplishment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.122, ANCOVA — P-Value for Role Performance; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.931, ANCOVA — P-Value for Communication; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.788, ANCOVA — P-Value for Affective Expression; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.190, ANCOVA — P-Value for Involvement; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.360, ANCOVA — P-Value for Control; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.446, ANCOVA — P-Value for Values and Norms; Model included treatment, pooled investigator, child with ADHD, and baseline

4. Secondary Outcome: Change From Baseline to 8 Weeks in the Family Assessment Measure Version III (FAM) Dyadic Relationship Scale (DRS) - Spouse/Significant Other
Description: FAM consists of 3 components: General Scale; Dyadic Relationships Scale (DRS), and Self-Rating Scale. The spouse/significant other completed the DRS scale, a 42-item self-report scale providing quantitative indices of family strengths/weaknesses. Items are rated 0-3 (strongly agree, agree, disagree, strongly disagree). Raw scores=0-18 (each subscale) and are converted to a t-score (mean=50, standard deviation (SD)=10; scores range from 0-100). T-scores should be between 40-60. T-scores >=60 indicate disturbance in family functioning.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-scores of units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
T-scores of units on a scale
  Task Accomplishment | -0.28 (6.57) | 0.15 (7.10)
  Role Performance | -0.86 (5.86) | -0.35 (6.33)
  Communication | -0.15 (7.24) | -0.05 (7.21)
  Affective Expression | 0.17 (8.30) | 0.32 (8.83)
  Involvement | -0.25 (7.50) | 0.11 (7.81)
  Control | 0.15 (6.46) | 0.54 (6.78)
  Values and Norms | -0.27 (8.15) | -0.95 (7.08)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.575, ANCOVA — P-Value for Task Accomplishment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.705, ANCOVA — P-Value for Role Performance; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.686, ANCOVA — P-Value for Communication; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.618, ANCOVA — P-Value for Affective Expression; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.903, ANCOVA — P-Value for Involvement; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.807, ANCOVA — P-Value for Control; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.403, ANCOVA — P-Value for Values and Norms; Model included treatment, pooled investigator, child with ADHD, and baseline

5. Secondary Outcome: Change From Baseline to 24 Weeks in the Family Assessment Measure Version III (FAM) Dyadic Relationship Scale (DRS) - Spouse/Significant Other
Description: as for outcome 4
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-scores of units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
T-scores of units on a scale
  Task Accomplishment | -0.79 (6.94) | 0.24 (6.99)
  Role Performance | -0.93 (6.03) | -0.41 (6.37)
  Communication | 0.14 (7.09) | -0.09 (7.17)
  Affective Expression | -0.08 (8.02) | 0.60 (8.79)
  Involvement | -0.47 (7.88) | -0.10 (7.69)
  Control | 0.05 (7.15) | 0.73 (6.69)
  Values and Norms | -0.19 (8.00) | -0.57 (7.34)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.941, ANCOVA — P-Value for Task Accomplishment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.788, ANCOVA — P-Value for Role Performance; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.391, ANCOVA — P-Value for Communication; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.685, ANCOVA — P-Value for Affective Expression; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.774, ANCOVA — P-Value for Involvement; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.360, ANCOVA — P-Value for Control; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.446, ANCOVA — P-Value for Values and Norms; Model included treatment, pooled investigator, child with ADHD, and baseline

6. Secondary Outcome: Change From Baseline to 8 Weeks in the Dyadic Adjustment Scale (DAS) - Participant
Description: 32-item self-report scale to assess quality of the relationship perceived by participants. Response anchors vary and include a 5-, 6- or 7-point Likert scale (always agree/disagree; all the time/never); and 2 yes/no items. Assesses 4 relationship aspects (# items): dyadic satisfaction (10), cohesion (5), consensus (13), affectional expression (4). Raw score total=0-151 and is converted to a t-score (0-100; mean=50, standard deviation (SD)=10). T-scores of 45-55 indicate a typical score (no concern). Scores <30 indicate significant impairment. Lower scores indicate poorer dyadic adjustment.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-scores of units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
T-scores of units on a scale
  Total Dyadic Adjustment | 1.13 (6.33) | 0.70 (6.55)
  Dyadic Consensus | 1.61 (6.77) | 1.42 (7.22)
  Dyadic Satisfaction | 0.52 (6.22) | -0.02 (5.53)
  Affectional Expression | 1.16 (9.00) | -0.85 (8.27)
  Dyadic Cohesion | -0.06 (7.65) | 0.54 (6.86)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.617, ANCOVA — P-Value for Total Dyadic Adjustment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.789, ANCOVA — P-Value for Dyadic Consensus; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.670, ANCOVA — P-Value for Dyadic Satisfaction; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.018, ANCOVA — P-Value for Affectional Expression; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.405, ANCOVA — P-Value for Dyadic Cohesion; Model included treatment, pooled investigator, child with ADHD, and baseline

7. Secondary Outcome: Change From Baseline to 24 Weeks in the Dyadic Adjustment Scale (DAS) - Participant
Description: 32-item self-report scale to assess quality of the relationship perceived by participants. Response anchors vary and include a 5-, 6- or 7-point Likert scale (always agree/disagree; all the time/never); and 2 yes/no items. Assesses 4 relationship aspects (# items): dyadic satisfaction (10), cohesion (5), and consensus (13), and affectional expression (4). Raw score total=0-151 and is converted to a t-score (0-100; mean=50, SD=10). T-scores of 45-55 indicate a typical score (no concern). Scores <30 indicate significant impairment. Lower scores indicate poorer dyadic adjustment.
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-scores of units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
T-scores of units on a scale
  Total Dyadic Adjustment | 1.21 (7.12) | 0.51 (7.74)
  Dyadic Consensus | 2.13 (6.97) | 1.58 (8.34)
  Dyadic Satisfaction | 0.47 (6.83) | -0.32 (6.13)
  Affectional Expression | 0.62 (9.09) | -1.13 (9.93)
  Dyadic Cohesion | 0.30 (7.92) | 0.16 (8.01)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.544, ANCOVA — P-Value for Total Dyadic Adjustment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.494, ANCOVA — P-Value for Dyadic Consensus; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.547, ANCOVA — P-Value for Dyadic Satisfaction; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.059, ANCOVA — P-Value for Affectional Expression; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.918, ANCOVA — P-Value for Dyadic Cohesion; Model included treatment, pooled investigator, child with ADHD, and baseline

8. Secondary Outcome: Change From Baseline to 8 Weeks in the Dyadic Adjustment Scale (DAS) - Spouse/Significant Other
Description: 32-item self-report scale to assess quality of the relationship perceived by the spouse/significant other. Response anchors vary and include a 5-, 6- or 7-point Likert scale (always agree/disagree; all the time/never); and 2 yes/no items. Assesses 4 relationship aspects (# items): dyadic satisfaction (10), cohesion (5), and consensus (13), and affectional expression (4). Raw score total=0-151 and is converted to a t-score (0-100; mean=50, SD=10). T-scores of 45-55 indicate a typical score (no concern). Scores <30 indicate significant impairment. Lower scores indicate poorer dyadic adjustment.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-scores of units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 246 | 215
T-scores of units on a scale
  Total Dyadic Adjustment | 2.09 (6.37) | 2.64 (7.13)
  Dyadic Consensus | 2.49 (6.84) | 3.67 (7.92)
  Dyadic Satisfaction | 1.37 (5.81) | 1.61 (6.36)
  Affectional Expression | 1.57 (9.40) | 1.23 (9.57)
  Dyadic Cohesion | 0.81 (7.33) | 0.29 (8.23)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.334, ANCOVA — P-Value for Total Dyadic Adjustment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.087, ANCOVA — P-Value for Dyadic Consensus; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.795, ANCOVA — P-Value for Dyadic Satisfaction; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.955, ANCOVA — P-Value for Affectional Expression; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.788, ANCOVA — P-Value for Dyadic Cohesion; Model included treatment, pooled investigator, child with ADHD, and baseline

9. Secondary Outcome: Change From Baseline to 24 Weeks in the Dyadic Adjustment Scale (DAS) - Spouse/Significant Other
Description: as for outcome 8
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-scores of units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 246 | 215
T-scores of units on a scale
  Total Dyadic Adjustment | 2.09 (6.97) | 2.84 (6.80)
  Dyadic Consensus | 2.79 (7.49) | 3.87 (7.22)
  Dyadic Satisfaction | 1.32 (6.17) | 1.27 (6.47)
  Affectional Expression | 1.38 (10.08) | 2.00 (8.00)
  Dyadic Cohesion | 0.87 (7.70) | 0.99 (7.60)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.248, ANCOVA — P-Value for Total Dyadic Adjustment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.163, ANCOVA — P-Value for Dyadic Consensus; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.947, ANCOVA — P-Value for Dyadic Satisfaction; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.214, ANCOVA — P-Value for Affectional Expression; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.543, ANCOVA — P-Value for Dyadic Cohesion; Model included treatment, pooled investigator, child with ADHD, and baseline

10. Primary Outcome: Change From Baseline to 12 Weeks in the Conners' Adult Attention Deficit Hyperactivity Disorder Rating Scale - Investigator Rated: Screening Version (CAARS-Inv:SV) Total ADHD Symptoms Score
Description: as for outcome 1
Time Frame: Baseline, 12 weeks
Population: Participants with a baseline and at least one post-baseline CAARS Total ADHD Symptoms Score were included. The protocol was amended to extend the open-label portion of the study from 8 weeks to 12 weeks, and the primary objective was modified to include the CAARS-IV:SV at 12 weeks.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 180 | 165
Units on a scale | -14.33 (0.83) | -10.05 (0.82)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Model included visit, baseline, treatment, pooled investigator, child with ADHD, and treatment by visit; Mean Difference (Final Values) = -4.28, Standard Error of Mean 1.05 — Least Squares Mean Difference = Atomoxetine - Placebo

11. Secondary Outcome: Change From Baseline to 8 Weeks in the Parenting Stress Index (PSI) Score - Total Stress and Life Stress
Description: The PSI 19-item Stress Life Events scale has yes/no responses and measures situational circumstances beyond control (death of family member, divorce, etc.) in the past 12 months. Maximum score (all answers=yes) is 79; a Life Stress raw score >=17 indicates high stress. Each question is weighted based upon the event. Total Score measures relative magnitude of stress in parent-child system. High scores (>=85th percentile) indicate higher stress. Total Stress >=258 is indicative of impairment. Participants with a child aged 6-12 or 13-17 years living at home completed the scale.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
Units on a scale
  Total Stress | -10.74 (32.14) | -7.06 (26.63)
  Life Stress | 0.25 (4.22) | -0.30 (4.04)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.446, ANCOVA — P-Value for Total Stress; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.134, ANCOVA — P-Value for Life Stress; Model included treatment, pooled investigator, child with ADHD, and baseline

12. Secondary Outcome: Change From Baseline to 8 Weeks in the Parenting Stress Index (PSI) Score - Parent Domains
Description: 120-item scale includes 101 items rated on 5-point Likert scale (strongly agree/strongly disagree) or 4-5 point multiple choices. Adult Domain characteristics' subscales and score ranges include: Competence (13-65), Isolation (6-30), Attachment (7-35), Health (5-25), Role Restriction (7-35), Depression (9-45), Spouse (7-35). Total Score measures relative magnitude of stress in parent-child system. Parent Domain score >=148 (>=85th percentile) is indicative of impairment. Participants with a child aged 6-12 or 13-17 years living at home completed the scale.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
Units on a scale
  Parent Domain Total | -5.08 (17.40) | -1.34 (12.95)
  Parent Domain Competence | -1.78 (5.29) | -1.24 (4.26)
  Parent Domain Isolation | -0.68 (3.55) | -0.11 (2.97)
  Parent Domain Attachment | 0.05 (3.34) | 0.40 (2.74)
  Parent Domain Health | 0.05 (2.48) | -0.05 (2.18)
  Parent Domain Role Restriction | -0.51 (4.07) | 0.06 (3.75)
  Parent Domain Depression | -1.55 (4.70) | -0.08 (3.78)
  Parent Domain Spouse | -0.74 (3.63) | -0.32 (3.72)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.056, ANCOVA — P-Value for Parent Domain Total; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.459, ANCOVA — P-Value for Parent Domain Competence; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.435, ANCOVA — P-Value for Parent Domain Isolation; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.677, ANCOVA — P-Value for Parent Domain Attachment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.376, ANCOVA — P-Value for Parent Domain Health; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.176, ANCOVA — P-Value for Parent Domain Role Restriction; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.030, ANCOVA — P-Value for Parent Domain Depression; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 8: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.434, ANCOVA — P-Value for Parent Domain Spouse; Model included treatment, pooled investigator, child with ADHD, and baseline

13. Secondary Outcome: Change From Baseline to 8 Weeks in the Parenting Stress Index (PSI) Score - Child Domains
Description: 120-item scale includes 101 items rated on 5-point Likert scale (strongly agree/strongly disagree) or 4-5 point multiple choices. Child Domain characteristics' subscales and score ranges include: Distractibility/Hyperactivity (9-45), Adaptability (11-55), Reinforces Parent (6-30), Demandingness (9-45), Mood (5-25), Acceptability (7-35). Total Score measures relative magnitude of stress in parent-child system. A Child Domain score >=116 (>=85th percentile) is indicative of impairment. Participants with a child aged 6-12 or 13-17 years living at home completed the scale.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
Units on a scale
  Child Domain Total | -5.66 (19.12) | -5.72 (18.62)
  Defensive Responding | -1.66 (5.48) | -0.35 (4.75)
  Child Domain Distractibility/Hyperactive | -1.70 (4.15) | -1.93 (4.11)
  Child Domain Adaptability | -1.56 (6.92) | -1.87 (7.23)
  Child Domain Reinforces Parent | -0.79 (4.98) | -0.32 (4.44)
  Child Domain Demandingness | -0.56 (3.78) | -1.00 (3.99)
  Child Domain Mood | -0.36 (2.63) | -0.26 (2.67)
  Child Domain Acceptability | -0.68 (3.48) | -0.34 (3.31)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.578, ANCOVA — P-Value for Child Domain Total; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.062, ANCOVA — P-Value for Defensive Responding; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.567, ANCOVA — P-Value for Child Domain Distractibility/Hyperactive; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.383, ANCOVA — P-Value for Child Domain Adaptability; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.963, ANCOVA — P-Value for Child Domain Reinforces Parent; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.075, ANCOVA — P-Value for Child Domain Demandingness; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.854, ANCOVA — P-Value for Child Domain Mood; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 8: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.671, ANCOVA — P-Value for Child Domain Acceptability; Model included treatment, pooled investigator, child with ADHD, and baseline

14. Secondary Outcome: Change From Baseline to 24 Weeks in the Parenting Stress Index (PSI) Score - Total Stress and Life Stress
Description: as for outcome 11
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
Units on a scale
  Total Stress | -17.19 (40.19) | -10.97 (31.33)
  Life Stress | 0.99 (4.91) | 0.19 (4.93)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.280, ANCOVA — P-Value for Total Stress; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.34, ANCOVA — P-Value for Life Stress; Model included treatment, pooled investigator, child with ADHD, and baseline

15. Secondary Outcome: Change From Baseline to 24 Weeks in the Parenting Stress Index (PSI) Score - Parent Domains
Description: as for outcome 12
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
Units on a scale
  Parent Domain Total | -7.66 (21.45) | -3.12 (15.18)
  Parent Domain Competence | -2.58 (5.77) | -1.57 (4.54)
  Parent Domain Isolation | -1.08 (3.61) | -0.28 (3.17)
  Parent Domain Attachment | -0.19 (3.53) | -0.01 (2.57)
  Parent Domain Health | -0.09 (2.75) | 0.07 (2.45)
  Parent Domain Role Restriction | -0.52 (4.58) | -0.31 (4.00)
  Parent Domain Depression | -2.13 (5.29) | -0.54 (4.29)
  Parent Domain Spouse | -0.75 (4.22) | -0.48 (3.70)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.103, ANCOVA — P-Value for Parent Domain Total; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.182, ANCOVA — P-Value for Parent Domain Competence; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.161, ANCOVA — P-Value for Parent Domain Isolation; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.472, ANCOVA — P-Value for Parent Domain Attachment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.949, ANCOVA — P-Value for Parent Domain Health; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.848, ANCOVA — P-Value for Parent Domain Role Restriction; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.050, ANCOVA — P-Value for Parent Domain Depression; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 8: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.840, ANCOVA — P-Value for Parent Domain Spouse; Model included treatment, pooled investigator, child with ADHD, and baseline

16. Secondary Outcome: Change From Baseline to 24 Weeks in the Parenting Stress Index (PSI) Score - Child Domains
Description: as for outcome 13
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 262 | 227
Units on a scale
  Child Domain Total | -9.52 (22.92) | -7.85 (20.07)
  Defensive Responding | -2.28 (6.44) | -0.84 (5.20)
  Child Domain Distractibility/Hyperactive | -2.28 (4.24) | -2.60 (4.35)
  Child Domain Adaptability | -2.66 (7.95) | -2.44 (7.28)
  Child Domain Reinforces Parent | -1.54 (5.58) | -0.63 (4.96)
  Child Domain Demandingness | -1.06 (4.14) | -1.30 (4.19)
  Child Domain Mood | -0.72 (2.89) | -0.33 (3.02)
  Child Domain Acceptability | -0.91 (3.75) | -0.56 (3.51)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.785, ANCOVA — P-Value for Child Domain Total; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.081, ANCOVA — P-Value for Defensive Responding; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.518, ANCOVA — P-Value for Child Domain Distractibility/Hyperactive; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.883, ANCOVA — P-Value for Child Domain Adaptability; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.439, ANCOVA — P-Value for Child Domain Reinforces Parent; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.167, ANCOVA — P-Value for Child Domain Demandingness; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.381, ANCOVA — P-Value for Child Domain Mood; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 8: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.906, ANCOVA — P-Value for Child Domain Acceptability; Model included treatment, pooled investigator, child with ADHD, and baseline

17. Secondary Outcome: Change From Baseline to 12 Weeks in the Alabama Parenting Questionnaire (APQ) Parent Form
Description: 42-item scale, 3 subscales (z-scores [-2 to 2]): Dysfunctional/Negative/Positive Parenting. Each construct rated 1=never/5=always (# items): involvement (10), supervision (10), positive parenting (6), inconsistent discipline (6), other discipline (7), harsh discipline (3). Higher scores indicate impairment: dysfunctional/negative parenting composite; supervision, inconsistent discipline, harsh punishment, other discipline. Lower scores indicate impairment: positive parenting composite; positive parenting, involvement. Completed by participants with a child 6-12 or 13-17 years living at home.
Time Frame: Baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 230 | 192
Units on a scale
  Parent Involvement (n=230, 192) | 0.27 (3.96) | 0.67 (3.57)
  Parent Positive Parenting (n=230, 192) | 0.00 (2.59) | 0.36 (2.33)
  Parent Poor Supervision (n=229, 191) | -1.29 (3.39) | -1.17 (3.43)
  Parent Inconsistent Discipline (n=230, 192) | -1.07 (2.78) | -0.81 (2.59)
  Parent Corporal Punishment (n=230, 192) | -0.23 (1.36) | -0.21 (1.00)
  Parent Other Discipline Practice (n=230, 190) | -0.01 (2.51) | 0.00 (2.57)
  Dysfunctional Parenting Composite (n=229, 191) | -0.23 (0.77) | -0.26 (0.65)
  Negative Parenting Composite (n=229, 191) | -0.37 (0.79) | -0.32 (0.74)
  Positive Parenting Composite (n=230, 192) | 0.03 (0.72) | 0.13 (0.64)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.420, ANCOVA — P-Value for Parent Involvement; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.249, ANCOVA — P-Value for Parent Positive Parenting; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.927, ANCOVA — P-Value for Parent Poor Supervision; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.205, ANCOVA — P-Value for Parent Inconsistent Discipline; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.673, ANCOVA — P-Value for Parent Corporal Punishment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.881, ANCOVA — P-Value for Parent Other Discipline Practice; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.808, ANCOVA — P-Value for Dysfunctional Parenting Composite; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 8: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.498, ANCOVA — P-Value for Negative Parenting Composite; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 9: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.283, ANCOVA — P-Value for Positive Parenting Composite; Model included treatment, pooled investigator, child with ADHD, and baseline

18. Secondary Outcome: Change From Baseline to 24 Weeks in the Alabama Parenting Questionnaire (APQ) Parent Form
Description: as for outcome 17
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 230 | 292
Units on a scale
  Parent Involvement (n=230, 192) | 0.31 (3.84) | 0.43 (3.47)
  Parent Positive Parenting (n=230, 192) | 0.07 (2.83) | 0.11 (2.35)
  Parent Poor Supervision (n=229, 191) | -1.24 (3.89) | -0.96 (3.31)
  Inconsistent Discipline (n=230, 192) | -1.19 (2.94) | -0.82 (2.75)
  Parent Corporal Punishment (n=230, 192) | -0.25 (1.34) | -0.14 (1.17)
  Other Discipline Practice (n=230, 190) | 0.22 (2.67) | 0.18 (2.27)
  Dysfunctional Parenting Composite (n=229, 191) | -0.25 (0.80) | -0.20 (0.56)
  Negative Parenting Composite (n=229, 191) | -0.39 (0.86) | -0.28 (0.71)
  Positive Parenting Composite (n=230, 192) | 0.05 (0.74) | 0.07 (0.61)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.784, ANCOVA — P-Value for Parent Involvement; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.864, ANCOVA — P-Value for Parent Positive Parenting; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.884, ANCOVA — P-Value for Parent Poor Supervision; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.072, ANCOVA — P-Value for Parent Inconsistent Discipline; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.120, ANCOVA — P-Value for Parent Corporal Punishment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.925, ANCOVA — P-Value Other Discipline Practice; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.444, ANCOVA — P-Value for Dysfunctional Parenting Composite; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 8: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.166, ANCOVA — P-Value for Negative Parenting Composite; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 9: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.875, ANCOVA — P-Value for Positive Parenting Composite; Model included treatment, pooled investigator, child with ADHD, and baseline

19. Secondary Outcome: Change From Baseline to 12 Weeks in the Alabama Parenting Questionnaire (APQ) Child Form
Description: 42-item scale, 3 subscales (z-scores [-2 to 2]): Dysfunctional/Negative/Positive Parenting. Each construct rated 1=never/5=always (# items): involvement (10), supervision (10), positive parenting (6), inconsistent discipline (6), other discipline (7), harsh discipline (3). Higher scores indicate impairment: dysfunctional/negative parenting composite; supervision, inconsistent discipline, harsh punishment, other discipline. Lower scores indicate impairment: positive parenting composite; positive parenting, involvement. Completed by child 6-12 or 13-17 years living at home.
Time Frame: Baseline, 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 189 | 159
Units on a scale
  Child Involvement Mother (n=189, 158) | 0.08 (5.40) | -0.17 (5.41)
  Child Involvement Father (n=188, 159) | 0.38 (5.89) | -0.15 (5.37)
  Child Positive Parenting (n=188, 159) | -0.80 (3.77) | -0.24 (3.98)
  Child Poor Supervision (n=188, 158) | -1.12 (4.44) | -1.23 (4.27)
  Child Inconsistent Discipline (n=189,159) | -0.60 (3.44) | -0.81 (3.67)
  Child Corporal Punishment (n=189, 160) | -0.30 (1.78) | -0.31 (1.66)
  Child Other Discipline Practice (n=189, 159) | -0.24 (3.71) | -0.27 (3.77)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.895, ANCOVA — P-Value for Child Involvement Mother; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.792, ANCOVA — P-Value for Child Involvement Father; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.318, ANCOVA — P-Value for Child Positive Parenting; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.914, ANCOVA — P-Value for Child Poor Supervision; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.961, ANCOVA — P-Value for Child Inconsistent Discipline; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.807, ANCOVA — P-Value for Child Corporal Punishment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.827, ANCOVA — P-Value for Child Other Discipline Practice; Model included treatment, pooled investigator, child with ADHD, and baseline

20. Secondary Outcome: Change From Baseline to 24 Weeks in the Alabama Parenting Questionnaire (APQ) Child Form
Description: as for outcome 19
Time Frame: Baseline, 24 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 189 | 160
Units on a scale
  Child Involvement Mother (n=189, 159) | 0.12 (5.94) | -0.11 (5.41)
  Child Involvement Father (n=188, 159) | 0.36 (6.25) | 0.44 (5.48)
  Child Positive Parenting (n=188, 159) | -0.90 (3.85) | -0.33 (4.05)
  Child Poor Supervision (n=188, 158) | -1.52 (4.60) | -1.31 (4.13)
  Child Inconsistent Discipline (n=189, 159) | -0.44 (3.61) | -0.86 (3.73)
  Child Corporal Punishment (n=189, 160) | -0.25 (1.99) | -0.34 (1.95)
  Child Other Discipline Practice (n=189, 159) | -0.24 (3.97) | -0.19 (4.02)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.828, ANCOVA — P-Value for Child Involvement Mother; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.401, ANCOVA — P-Value for Child Involvement Father; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.300, ANCOVA — P-Value for Child Positive Parenting; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.575, ANCOVA — P-Value for Child Poor Supervision; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.772, ANCOVA — P-Value for Child Inconsistent Discipline; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.918, ANCOVA — P-Value for Child Corporal Punishment; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.636, ANCOVA — P-Value for Child Other Discipline Practice; Model included treatment, pooled investigator, child with ADHD, and baseline

21. Secondary Outcome: Mean Change From Baseline to 24 Weeks in the Child Disruptive Behavior Rating Scale (CDBRS) Parent Form
Description: Contains the symptoms of ADHD (9 items for Inattention/9 items for Hyperactive-Impulsive). Total maximum severity score is 54 (0-27 for each subscale). Higher scores indicate greater impairment. Participants with a child 6-12 years old living in the home completed the scale.
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 181 | 159
Units on a scale
  Total ADHD Score | -2.93 (8.58) | -2.57 (8.91)
  Hyperactive-Impulsive Symptom ADHD Score | -1.18 (4.43) | -1.26 (4.48)
  Inattention Symptom ADHD Score | -1.75 (4.98) | -1.30 (5.22)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.583, ANCOVA — P-Value for Total ADHD Score; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.997, ANCOVA — P-Value for Hyperactive-Impulsive Symptom ADHD Score; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.333, ANCOVA — P-Value for Inattention Symptom ADHD Score; Model included treatment, pooled investigator, child with ADHD, and baseline

22. Secondary Outcome: Mean Change From Baseline to 24 Weeks in the Child Disruptive Behavior Rating Scale (CDBRS) Parent Form Oppositional Defiant Disorder (ODD) and Conduct Disorder Flags
Description: Items 19-26 of the CDBRS assess the presence of Oppositional Defiant Disorder (ODD) (yes if participant answers >=4 items as 2 [often] or 3 [very often]). Items 1-26 are rated on a 0-3 scale (0=never/rarely, 1=sometimes, 2=often, 3=very often). 15 yes/no items assess the presence of Conduct Disorder (yes if >3 items answered yes). Participants with a child 6-12 years old living in the home completed the scale.
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 125 | 136
Participants
  ODD Flag - Yes, Baseline | 54 | 40
  ODD Flag -No, Baseline | 127 | 119
  ODD Flag - Yes, 24 Weeks | 40 | 33
  ODD Flag -No, 24 Weeks | 141 | 126
  Conduct Disorder Flag - Yes, Baseline | 13 | 14
  Conduct Disorder Flag - No, Baseline | 168 | 145
  Conduct Disorder Flag - Yes, 24 Weeks | 14 | 10
  Conduct Disorder Flag - No, 24 Weeks | 167 | 149
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = .792, Fisher Exact — P-Value for Oppositional Defiant Disorder Flag
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.675, Fisher Exact — P-Value for Conduct Disorder Flag

23. Secondary Outcome: Change From Baseline to 8 Weeks in the Parenting Sense of Competence (PSOC) Scale
Description: 16-item scale to assess parenting self-esteem: the Satisfaction Subscale has 9 questions (2,3,4,5,8,9,12,14,16)=54; the Efficacy Subscale has 7 questions (1,6,7,10,11,13,15)=43. Each response on the satisfaction subscale is answered on a 6-point scale (strongly agree/strongly disagree). Higher scores indicate greater satisfaction and greater self-efficacy. Lower scores mean more impairment. Participants with a child aged 6-12 or 13-17 years living at home completed the scale.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 261 | 227
Units on a scale
  Total Score | 3.51 (7.95) | 2.52 (6.44)
  Satisfaction Scale | 1.77 (5.63) | 1.26 (5.03)
  Efficacy Scale | 1.75 (3.80) | 1.25 (3.21)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.875, ANCOVA — P-Value for PSOC Total; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.569, ANCOVA — P-Value for Satisfaction Scale; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.399, ANCOVA — P-Value for Efficacy Scale; Model included treatment, pooled investigator, child with ADHD, and baseline

24. Secondary Outcome: Change From Baseline to 24 Weeks in the Parenting Sense of Competence (PSOC) Scale
Description: as for outcome 23
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 261 | 227
Units on a scale
  Total Score | 4.57 (8.57) | 2.93 (7.19)
  Satisfaction Scale | 2.48 (6.00) | 1.53 (5.60)
  Efficacy Scale | 2.09 (3.96) | 1.41 (3.32)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.365, ANCOVA — P-Value for PSOC Total; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.620, ANCOVA — P-Value for Satisfaction Scale; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.462, ANCOVA — P-Value for Efficacy Scale; Model included treatment, pooled investigator, child with ADHD, and baseline

25. Secondary Outcome: Change From Baseline to 12 and 24 Weeks in the Adult Attention Deficit Hyperactivity Disorder Investigator Symptom Rating Scale Total and Subscale Scores
Description: 18-item scale that captures the 18-item DSM-IV symptoms of ADHD. 9 inattentive items alternate with 9 hyperactive/impulsive items. Each item is scored 0 (none), 1 (mild), 2 (moderate), or 3 (severe). The total score range is 0-54 (0-27 for each subscale). Higher scores indicate more impaired participants. The scale was administered by a physician or PhD at the investigative site.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 235 | 202
Units on a scale
  Total Score 12 Weeks (n=233, 201) | -13.26 (11.95) | -9.06 (11.11)
  Hyperactivity Score 12 Weeks (n=233, 202) | -5.84 (6.18) | -4.37 (6.05)
  Inattention Score 12 Weeks (n=233, 201) | -7.42 (6.77) | -4.66 (6.44)
  Total Score 24 Weeks (n=235, 202) | -13.66 (12.54) | -8.02 (11.01)
  Hyperactivity Score 24 Weeks (n=235, 202) | -6.05 (6.55) | -3.68 (5.79)
  Inattention Score 24 Weeks (n=235, 202) | -7.62 (6.96) | -4.35 (6.26)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — P-Value for Total Score at 12 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA — P-Value for Hyperactivity Score at 12 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value for Inattention Score at 12 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value for Total Score at 24 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value for Hyperactivity Score at 24 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value for Inattention Score at 24 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline

26. Secondary Outcome: Change From Baseline to 8 and 24 Weeks in the Clinical Global Improvement Attention Deficit Hyperactivity Disorder Severity (CGI-ADHD-S)
Description: The CGI-ADHD-S is a single-item rating of the clinician's assessment of the severity of ADHD symptoms in relation to the clinician's total experience with ADHD subjects. Severity is rated on a 7-point scale (1=normal, not at all ill; 7=among the most extremely ill subjects). The scale was administered by a physician or PhD at the investigative site.
Time Frame: Baseline, 8 weeks, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 264 | 232
Units on a scale
  8 Weeks | -1.13 (1.08) | -0.69 (0.91)
  24 Weeks | -1.18 (1.18) | -0.67 (1.03)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value for 8 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value for 24 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline

27. Secondary Outcome: Change From Baseline to 12 and 24 Weeks in the Montgomery-Asberg Depression Rating Scale Total Score (MADRS)
Description: The MADRS is an investigator administered rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline 12 weeks, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 236 | 202
Units on a scale
  12 Weeks (n=235,202) | -0.69 (5.90) | 0.14 (6.25)
  24 Weeks (n=236,202) | -0.61 (6.53) | 0.36 (6.19)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.553, ANCOVA — P-Value for 12 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.797, ANCOVA — P-Value for 24 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline

28. Secondary Outcome: Change From Baseline to 12 and 24 Weeks in the State-Trait Anxiety Inventories (STAI)
Description: Self-report scale completed by the participant. Separate scales measure state (20 items) and trait (20 items) anxiety. The participant reports how they feel "right now at this moment" for state anxiety and how they "generally" feel for trait anxiety. The "state" items are scored as: 1 (not at all), 2 (somewhat true), 3 (moderately true), 4 (very true). The "trait" items are scored as: 1 (almost never), 2 (sometimes), 3 (often), 4 (almost always). Scores range from 4-80 for each scale. Higher scores indicate more impaired participants.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 233 | 198
Units on a scale
  State Anxiety Score 12 Weeks (n=230, 197) | -1.50 (11.96) | 1.12 (11.91)
  Trait Anxiety Score 12 Weeks (n=231, 198) | -5.67 (9.65) | -2.42 (9.29)
  State Anxiety Score 24 Weeks (n=232, 198) | -0.40 (13.22) | 0.38 (12.44)
  Trait Anxiety Score 24 Weeks (n=233, 198) | -5.32 (10.51) | -2.77 (9.60)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.108, ANCOVA — P-Value for State Anxiety Score at 12 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.026, ANCOVA — P-Value for Trait Anxiety Score at 12 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.897, ANCOVA — P-Value is for State Anxiety Score at 24 Weeks; Model included treatment, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine vs Placebo; Test type: Superiority or Other; p = 0.171, ANCOVA — P-Value is for Trait Anxiety Score at 24 weeks; Model included treatment, pooled investigator, child with ADHD, and baseline

29. Secondary Outcome: Change From Baseline to 1 Week of Titration in the CAARS-Inv:SV Total Attention Deficit Hyperactivity Disorder (ADHD) Symptoms and Subscale Scores
Description: as for outcome 1
Time Frame: Baseline, 1 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Atomoxetine Group 1: Atomoxetine 40 milligrams (mg)/day for 3 days followed by 80 mg/day for 4 days
- Atomoxetine Group 2: Atomoxetine 40 mg/day for 7 days followed by 80 mg/day for 7 days
- Placebo: Placebo is administered once daily, orally for 24 weeks. At the end of 24 weeks, the placebo arm is titrated to atomoxetine for 2 weeks then 40-100 mg/day
Arm/Group | Atomoxetine Group 1 | Atomoxetine Group 2 | Placebo
Number analyzed (Participants) | 144 | 119 | 232
Units on a scale
  Total ADHD Symptoms Score (n=144, 119) | -7.92 (8.51) | -7.62 (8.40) | -5.12 (8.34)
  Hyper/Impulsive Subscale (n=144, 119) | -3.21 (4.41) | -3.51 (4.39) | -2.41 (4.56)
  Inattention Subscale (n=144, 119) | -4.72 (5.28) | -4.11 (5.28) | -2.71 (4.78)
  ADHD Index Subscale (n=143, 119) | -4.65 (5.40) | -4.30 (5.59) | -2.53 (5.24)
Statistical Analysis 1: Comparison: Atomoxetine Group 1 vs Atomoxetine Group 2; Test type: Superiority or Other; p = 0.892, ANCOVA — P-Value for Total ADHD Symptoms Score; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine Group 1 vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — P-Value for Total ADHD Symptoms Score; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine Group 2 vs Placebo; Test type: Superiority or Other; p = 0.007, ANCOVA — P-Value for Total ADHD Symptoms Score; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine Group 1 vs Atomoxetine Group 2; Test type: Superiority or Other; p = 0.533, ANCOVA — P-Value for Hyper/Impulsive Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine Group 1 vs Placebo; Test type: Superiority or Other; p = 0.054, ANCOVA — P-Value for Hyper/Impulsive Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine Group 2 vs Placebo; Test type: Superiority or Other; p = 0.012, ANCOVA — P-Value for Hyper/Impulsive Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine Group 1 vs Atomoxetine Group 2; Test type: Superiority or Other; p = 0.457, ANCOVA — P-Value for Inattention Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 8: Comparison: Atomoxetine Group 1 vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA — P-Value for Inattention Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 9: Comparison: Atomoxetine Group 2 vs Placebo; Test type: Superiority or Other; p = 0.021, ANCOVA — P-Value for Inattention Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 10: Comparison: Atomoxetine Group 1 vs Atomoxetine Group 2; Test type: Superiority or Other; p = 0.710, ANCOVA — P-Value for ADHD Index Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 11: Comparison: Atomoxetine Group 1 vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — P-Value for ADHD Index Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 12: Comparison: Atomoxetine Group 2 vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA — P-Value for ADHD Index Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline

30. Secondary Outcome: Change From Baseline to 2 Weeks of Titration in the CAARS-Inv:SV Total Attention Deficit Hyperactivity Disorder (ADHD) Symptoms and Subscale Scores
Description: as for outcome 1
Time Frame: Baseline, 2 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Atomoxetine Group 1: Atomoxetine 40 milligrams (mg)/day for 3 days followed by 80 mg/day for 11 days
Arm/Group | Atomoxetine Group 1 | Atomoxetine Group 2 | Placebo
Number analyzed (Participants) | 144 | 119 | 232
Units on a scale
  Total ADHD Symptoms Score | -10.55 (9.41) | -10.58 (10.24) | -7.77 (9.38)
  Hyper/Impulsive Subscale | -4.61 (4.53) | -4.76 (5.15) | -3.43 (5.02)
  Inattention Subscale | -5.94 (5.83) | -5.83 (6.39) | -4.34 (5.51)
  ADHD Index Subscale | -6.09 (6.11) | -5.92 (6.61) | -4.00 (5.70)
Statistical Analysis 1: Comparison: Atomoxetine Group 1 vs Atomoxetine Group 2; Test type: Superiority or Other; p = 0.722, ANCOVA — P-Value for Total ADHD Symptoms Score; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Atomoxetine Group 1 vs Placebo; Test type: Superiority or Other; p = 0.011, ANCOVA — P-Value for Total ADHD Symptoms Score; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Atomoxetine Group 2 vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA — P-Value for Total ADHD Symptoms Score; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Atomoxetine Group 1 vs Atomoxetine Group 2; Test type: Superiority or Other; p = 0.779, ANCOVA — P-Value for Hyper/Impulsive Scale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 5: Comparison: Atomoxetine Group 1 vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA — P-Value for Hyper/Impulsive Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 6: Comparison: Atomoxetine Group 2 vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — P-Value for Hyper/Impulsive Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 7: Comparison: Atomoxetine Group 1 vs Atomoxetine Group 2; Test type: Superiority or Other; p = 0.716, ANCOVA — P-Value for Inattention Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 8: Comparison: Atomoxetine Group 1 vs Placebo; Test type: Superiority or Other; p = 0.071, ANCOVA — P-Value for Inattention Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 9: Comparison: Atomoxetine Group 2 vs Placebo; Test type: Superiority or Other; p = 0.034, ANCOVA — P-Value for Inattention Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 10: Comparison: Atomoxetine Group 1 vs Atomoxetine Group 2; Test type: Superiority or Other; p = 0.938, ANCOVA — P-Value for ADHD Index Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 11: Comparison: Atomoxetine Group 1 vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA — P-Value for ADHD Index Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 12: Comparison: Atomoxetine Group 2 vs Placebo; Test type: Superiority or Other; p = 0.005, ANCOVA — P-Value for ADHD Index Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline

31. Secondary Outcome: Change From Baseline to After a 2-Week Titration Period Beginning at Week 24 and Ending at Week 26 in the CAARS-Inv:SV Total Attention Deficit Hyperactivity Disorder (ADHD) Symptoms and Subscale Scores: Dosing Titration Strategy After Placebo
Description: as for outcome 1
Time Frame: Baseline, after 2-week titration period beginning at Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo/Atomoxetine Group 1: Placebo for 24 Weeks followed by atomoxetine 40 milligrams (mg)/day for 3 days followed by 80 mg/day for 11 days
- Placebo/Atomoxetine Group 2: Placebo for 24 weeks followed by atomoxetine 40 mg/day for 7 days followed by 80 mg/day for 7 days
- Atomoxetine: Atomoxetine for 24 weeks
Arm/Group | Placebo/Atomoxetine Group 1 | Placebo/Atomoxetine Group 2 | Atomoxetine
Number analyzed (Participants) | 67 | 66 | 119
Units on a scale
  Total ADHD Symptoms Score | -4.54 (7.23) | -4.92 (9.67) | -0.17 (5.89)
  Hyper/Impulsive Subscale | -1.71 (4.28) | -2.00 (4.71) | -0.06 (2.75)
  Inattention Subscale | -2.82 (4.32) | -2.92 (5.59) | -0.12 (3.79)
  ADHD Index Subscale | -2.37 (4.95) | -2.91 (6.72) | -0.17 (4.21)
Statistical Analysis 1: Comparison: Placebo/Atomoxetine Group 1 vs Placebo/Atomoxetine Group 2; Test type: Superiority or Other; p = 0.546, ANCOVA — P-Value for Total ADHD Symptoms Score; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 2: Comparison: Placebo/Atomoxetine Group 1 vs Placebo/Atomoxetine Group 2; Test type: Superiority or Other; p = 0.530, ANCOVA — P-Value for Hyper/Impulsive Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 3: Comparison: Placebo/Atomoxetine Group 1 vs Placebo/Atomoxetine Group 2; Test type: Superiority or Other; p = 0.569, ANCOVA — P-Value for Inattention Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline
Statistical Analysis 4: Comparison: Placebo/Atomoxetine Group 1 vs Placebo/Atomoxetine Group 2; Test type: Superiority or Other; p = 0.986, ANCOVA — P-Vaue for ADHD Index Subscale; Model included visit by therapy, pooled investigator, child with ADHD, and baseline

ADVERSE EVENTS:
Description: 266 participants received study drug and were included in the safety analyses.
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 4/266 | 3/234
Other Adverse Events (participants affected / at risk) | 248/266 | 191/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=266) | Placebo (N=234)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=266) | Placebo (N=234)
Abdominal pain upper (Gastrointestinal disorders) | 14 (15) | 2 (2)
Constipation (Gastrointestinal disorders) | 17 (19) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 69 (73) | 11 (11)
Nausea (Gastrointestinal disorders) | 91 (110) | 17 (20)
Vomiting (Gastrointestinal disorders) | 15 (15) | 6 (6)
Fatigue (General disorders) | 38 (43) | 20 (20)
Irritability (General disorders) | 25 (28) | 19 (21)
Nasopharyngitis (Infections and infestations) | 14 (15) | 29 (29)
Sinusitis (Infections and infestations) | 14 (15) | 9 (11)
Upper respiratory tract infection (Infections and infestations) | 13 (13) | 13 (15)
Decreased appetite (Metabolism and nutrition disorders) | 53 (55) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 14 (14)
Dizziness (Nervous system disorders) | 30 (34) | 11 (11)
Headache (Nervous system disorders) | 57 (68) | 62 (79)
Paraesthesia (Nervous system disorders) | 19 (19) | 2 (2)
Somnolence (Nervous system disorders) | 23 (24) | 9 (9)
Insomnia (Psychiatric disorders) | 35 (38) | 13 (13)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 16 (19) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days